CLINICAL TRIAL: NCT02586480
Title: Evolution of the PR Interval in Patients Implanted With a Dual Chamber Pacemaker With Algorithm for Spontaneous AV Conduction Preservation
Brief Title: Evolution of the PR Interval in Patients Implanted With a Pacemaker Using the SafeR Mode
Acronym: PRECISE
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: RBSY02
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Sinus Node Dysfunction; Atrioventricular Block
Keywords: bradycardia
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: dual chamber pacemaker with SafeR algorithm — SafeR is an AVB management algorithm: it provides AAI pacing while continuously monitoring AV conduction, it switches to DDD when detecting AVB I, II or III, according to the following criteria: (1) AVB I: 6 long PR intervals, (2) AVB II: 3 blocked atrial events/12 cycles, (3) AVB III: 2 consecutive blocked atrial events. It switches back to AAI mode when needed.
  Other Names: Reply DR (Sorin Devices)

SUMMARY:
Observational study on long PR interval using the SafeR mode in bradycardia patients.

DETAILED DESCRIPTION:
This observational trial aims to study the evolution of the PR interval in patients implanted with a dual chamber pacemaker with the SafeR mode. The investigators will assess the prevalence and the incidence of PR lengthening and the investigators will study the long PR interval management by physicians, depending on the data embedded in the pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted (primo-implant, replacement, upgrade) with a Sorin Group™ dual chamber pacemaker according to current available guidelines and IFU from less than three months.
* Since implantation, the device is programmed in SafeR mode
* Patient agreed to participate, after having received the appropriate and mandatory information

Exclusion Criteria:

* Patient contraindicated for cardiac pacing, according to current available guidelines
* Permanent atrial fibrillation
* Permanent high-degree AV block
* Patient not available for routine follow-up visits
* Patient already included in another clinical study
* Inability to understand the purpose of the study / refusal to cooperate
* minor age
* Pregnancy
* Life expectancy less than 12 months
* Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bradycardia patients eligible for dual chamber pacemaker implantation for SND, AVBI or AVBII
Sampling Method: Non-Probability Sample
Enrollment: 848 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prolonged PR interval (> 200ms) in patients without AVB I at baseline (Incidence of "clinical" AVB1) | at 12 months
  This incidence will be measured using PR/AR histograms stored in the device memory

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme TAIEB, MD, Principal Investigator — CH du Pays d'Aix - Aix en Provence
Locations (58):
- France (58):
  - CH Basse Terre, Terre Basse, Guadeloupe
  - CH du Pays d'Aix, Aix-en-Provence
  - CH Alençon, Alençon
  - Cabinet Alès, Alès
  - hôpital Sud, Amiens
  - CH Annecy, Annecy
  - hôpital privé Antony, Antony
  - hôpital d'Argenteuil, Argenteuil
  - hôpital St André, Bordeaux
  - CH Bourges, Bourges
  - CHU Brest, Brest
  - Clinique Keraudren, Brest
  - CHU Caen, Caen
  - Clinique des 2 Caps, Calais
  - CH Chartres, Chartres
  - Ch Chaumont, Chaumont
  - Cabinet Cherbourg, Cherbourg
  - HIA Percy, Clamart
  - Hôpital L. Pasteur, Colmar
  - CH Corbeil Essonnes, Corbeil-Essonnes
  - Cabinet Creutzwald, Creutzwald
  - Hopital Henri Mondor, Créteil
  - CH Dinan, Dinan
  - CH Douarnenez, Douarnenez
  - CH Evreux, Évreux
  - CMCO Evry, Évry
  - Cabinet Forbach, Forbach
  - CH Forbach, Forbach
  - CH Haguenau, Haguenau
  - CH Helfaut, Helfaut
  - CH Lannion, Lannion
  - CH Le Havre, Le Havre
  - CMCM Le Mans, Le Mans
  - CMC Port Marly, Le Port-Marly
  - CH Lomme, Lomme
  - CH Lorient, Lorient
  - CHU La Timone, Marseille
  - Hôpital Nord, Marseille
  - Clinique Melun, Melun
  - CH Privé Metz, Metz
  - CH Montfermeil, Montfermeil
  - Clinique Montpellier, Montpellier
  - Clinique A. Paré, Nancy
  - NCN Nantes, Nantes
  - CH Orléans, Orléans
  - Cabinet Paris, Paris
  - CH St Joseph, Paris
  - CH Poissy St Germain, Poissy
  - CHU Poitiers, Poitiers
  - Clinique St Hilaire, Rouen
  - CCN St Denis, Saint-Denis
  - CH St Nazaire, Saint-Nazaire
  - CH Sens, Sens
  - CH St Malo, St-Malo
  - CH Thionville, Thionville
  - CH Valenciennes, Valenciennes
  - Cabinet Valognes, Valognes
  - CH Villefrance, Villefranche-sur-Saône